CLINICAL TRIAL: NCT00079690
Title: Genetic Epidemiology of Blood Pressure Intervention
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1244; U01HL072507 (NIH)
Record Dates: First submitted 2004-03-10; First posted 2004-03-15 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2009-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To localize and identify new genes related to variation in blood pressure (BP) responses to a low dietary sodium intake, a high dietary sodium intake, oral potassium supplementation, and the cold pressor test.

DETAILED DESCRIPTION:
BACKGROUND:

Systemic hypertension is a complex disease determined by both genetic and environmental factors and is of significant public health interest. In addition, identifying genes that interact significantly with dietary sodium and potassium intake, or even the cold pressure test may enable clinicians to target life style modification for prevention and treatment of hypertension.

The study is conducted in response to a Request for Applications issued in October, 2001 on the Interaction of Genes and the Environment in Shaping Risk Factors for Heart, Lung, Blood, and Sleep Disorders.

DESIGN NARRATIVE:

The study uses a family intervention study design. The investigators will recruit 750 sibships (n=1750 siblings) and their parents (n=1250) from 500 families, each family ascertained through a proband who has untreated high normal BP or stage-1 hypertension (systolic BP 130-160 mm Hg and diastolic BP 85-100 mm Hg) from rural China. They will collect baseline information on medical history, lifestyle risk factors, anthropometric measures, BP, and blood measures (renin activity, ACE, angiotensin II, natriuretic peptide, glucose, insulin, and lipids) in all participants, and dietary nutrient intake (three 24-hour recalls) and urinary sodium and potassium excretion (three 24-hour) in the siblings. They will conduct the following interventions in the siblings: a cold pressor test at baseline (day 2 or 3), a 1-week low sodium-feeding study (40 mmol sodium/day on days 4-10), a 1-week high sodium-feeding study (280 mmol sodium/day on days 11-17), and a 1-week oral potassium supplementation (90 mmol potassium/day on days 18-24). They will measure BP and 24-hour urinary sodium and potassium excretion during the last 3 days of each intervention period. They will also perform genotyping for genomewide linkage scans and for candidate genes in all siblings and their parents. BP responses to the interventions will be analyzed primarily as quantitative traits. The primary analyses include linkage analysis, transmission/disequilibrium test, and association analysis between genetic markers and BP responses to the interventions.

ELIGIBILITY:
No eligibility criteria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2002-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiang He — Tulane University of Louisiana

REFERENCES:
- [Background] Huang J, Wildman RP, Gu D, Muntner P, Su S, He J. Prevalence of isolated systolic and isolated diastolic hypertension subtypes in China. Am J Hypertens. 2004 Oct;17(10):955-62. doi: 10.1016/j.amjhyper.2004.06.007. PMID 15485760
- [Background] Wildman RP, Gu D, Muntner P, Huang G, Chen J, Duan X, He J. Alcohol intake and hypertension subtypes in Chinese men. J Hypertens. 2005 Apr;23(4):737-43. doi: 10.1097/01.hjh.0000163141.82212.5f. PMID 15775777